CLINICAL TRIAL: NCT04711993
Title: Investigation of the Effects of Different Exercise Programs on Symptoms, Sleep, Cognitive Functions, Fatigue, Quality of Life, and Psychological Status in Patients With Restless Legs Syndrome.
Brief Title: Investigation of the Effects of Different Exercise Programs in Patients With Restless Legs Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Investigation of the effects of different exercise programs on symptoms, sleep, cognitive functions, fatigue, quality of life, and psychological status in patients with restless legs syndrome., Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-422.
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Restless Legs Syndrome; Anxiety; Sleep
MeSH Terms: conditions — Restless Legs Syndrome; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No application will be made to the control group. However, these patients will be included in the exercise program they want after the 8-week treatment period is completed.
- Aerobic exercise group (Experimental): Patients in the aerobic exercise group will exercise under the supervision of the therapist.
  Interventions: Other: Aerobic exercise
- Stretching exercise group (Experimental): Patients in the stretching-mobility exercise group will do stretching exercises under the supervision of the therapist
  Interventions: Other: Stretchin exercise

INTERVENTIONS:
Other: Aerobic exercise — Patients will do aerobic exercise three days a week for 40 minutes during 8 weeks. Aerobic exercise protocol will consist of warm up, loading and cooling periods. . Exercise prescription will be prepared in line with the recommendations of "The American College of Sports Medicine".
  Arms: Aerobic exercise group
Other: Stretchin exercise — Patients will do stretching exercise three days a week for 40 minutes during 8 weeks. Stretching exercises will start with active warm-up activities. Static stretching method will be used.
  Arms: Stretching exercise group

SUMMARY:
Restless leg syndrome (RLS) is a very common neurological condition characterized by an uncontrollable desire to move the legs. Due to the traumatic effect of RLS on morbidity, the patient is negatively affected in many different directions. The duration and quality of sleep of the patients decrease, and their cognitive functions change. The prevalence or risk of anxiety and depression increases in this population. At the same time, the quality of life of patients is significantly reduced. Among the different pharmacological agents used in RLS, dopamine agonists are the most widely used. However, the reporting of serious and common side effects related to this treatment has led to non-pharmacological approaches in the treatment of RLS and the effectiveness of many different approaches has been investigated. The exercise approach, which is determined to be effective in the treatment of the disease, is a subject that has been little studied. The type, duration and frequency of optimal exercise could not be standardized. In addition, the effect of exercise on RLS patients has been investigated in limited subjects. For this reason, the aim of our study is to examine the effect of different exercise programs on symptoms, sleep, cognitive functions, quality of life, psychological status and fatigue in patients with RLS.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with RLS according to the International Restless Legs Syndrome Study Group 2014 criteria
* Being over the age of 18
* Being literate
* Not having received any treatment for RLS, discontinuing treatment, or continuing symptoms despite current treatment.

Exclusion Criteria:

* Having any of musculoskeletal disorders that prevent physical activity
* History of ischemic heart disease (recent myocardial infarction or unstable angina, uncontrolled hypertension)
* Liver dysfunction
* Kidney dysfunction
* Anemia
* Diagnosis of another sleep disorder
* Diagnosis of gastrointestinal disease (irritable bowel syndrome, Crohn's disease, ulcerative colitis etc.)
* Pregnancy
* History of psychiatric, psychoactive, antidepressant medication use
* History of malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Symptoms | Before treatment, after treatment (end of 8 weeks)
  The severity of the symptoms of the patients will be evaluated with the International Restless Legs Syndrome Study Group Rating Scale. It is a 10-item questionnaire developed through expert evaluation of potential items. Scoring varies between 0-40. The higher the score indicates higher symptoms.
Change in Sleep | Before treatment, after treatment (end of 8 weeks)
  the patient will be asked to sleep by wearing watches that detect movement (movement watch) for 3 nights, one of which is fixed on the metatarsal and the other is fixed on the wrist. While the objective test of sleep is performed with the software compatible with the wrist watch, periodic extremity movements will be recorded with the software compatible with the other watch.
Change in Sleepiness | Before treatment, after treatment (end of 8 weeks)
  Epworth Sleepiness Scale(ESS) will be used. Its score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime
Change in Sleep Quality | Before treatment, after treatment (end of 8 weeks)
  Pittsburgh Sleep Quality Index will be used.Pittsburgh Sleep Quality Index scale has seven sub-scales that portray various domains of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Responses for each subscale are scored as 0-3. Having a global score of 5 or higher indicates bad sleep quality. sleepiness.

SECONDARY OUTCOMES:
Change in Psychological status | Before treatment, after treatment (end of 8 weeks)
  Psychological status of the patients will be evaluated with the Hospital Anxiety and Depression Scale. The scale has 14 items, 7 of which with odd numbers represent anxiety while the other 7 with even numbers represent depression. The scores range from 0 to 3 for each item and the maximum score in each sub-scale is 2. Higher scores means worse psychological status.
Change in Quality of life in RLS | Before treatment, after treatment (end of 8 weeks)
  Quality of life of the patients will be evaluated with the John Hopkins Restless Leg Syndrome Life Quality Questionnaire. It has 18 items. Ten of the items contribute to a single summary score, the overall life impact score. The remaining eight items concern employment (one question), sexual interest (two questions) and work (five questions).13 are scored on a 5-point scale which can be transformed to a 0-100 score, lower scores indicating worse quality of life. The remainder items are recorded as either a numerical value or a dichotomous response.
Change in Fatigue | Before treatment, after treatment (end of 8 weeks)
  Fatigue of the patients will be evaluated with the the Fatigue Severity Scale.The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Change in Gastrointestinal symptoms | Before treatment, after treatment (end of 8 weeks)
  Gastrointestinal symptoms of the patients will be evaluated with the Gastrointestinal Symptom Rating Scale.The GSRS is a 15-item 7-point Likert-type scale that evaluates how the individual feels in terms of GIS symptoms. It consists of five subcategories: abdominal pain, reflux, diarrhea, indigestion, and contipation. The 1st, 4th and 5th questions of the scale are about abdominal pain; 2. and 3. questions are about reflux; questions 11, 12 and 14 are about diarrhea; Questions 6, 7, 8, and 9 areabout indigestion; 10th, 13th and 15th questions are about constipation. Each item in the scale is valued between the statements of "no discomfort" and "very severe annoyance" and higher scores indicate that the symptoms are more severe.
Change in Cognitive function | Before treatment, after treatment (end of 8 weeks)
  Cognitive disfunction of the patients will be evaluated with the Cognitive Montreal Assessment Scale. Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Health Science Faculty, Ankara, Turkey (Türkiye)